CLINICAL TRIAL: NCT05943873
Title: Six Steps for a Successful Aesthetic Free Flap Reconstruction Shaping After Minimally Invasive Mastectomy
Brief Title: Successful Microsurgical Breast Reconstruction in Minimally Invasive Mastectomy
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Ju Huang, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 202300895B0
Record Dates: First submitted 2023-07-04; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Breast Reconstruction; Breast Cancer
Keywords: free flap; breast reconstruction; minimally invasive mastectomy; nipple-sparing mastectomy; robotic-assisted mastectomy; endoscopic-assisted mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Conventional mastectomy
- Minimally invasive: robotic-assisted or endoscopic assisted mastectomies

SUMMARY:
A retrospective chart review will be conducted to identify patients who received breast reconstruction surgery with DIEP flaps by a single plastic surgeon in one medical center between November 2018 and July 2022. Patients will be grouped based on how the mastectomy was performed, via minimally invasive or conventional approach. Demographic data, flap profile, vessel anastomosis and post-operative complication will be retrospectively reviewed. Data collection includes patient demographics, previous breast surgical history, breast cancer history and adjuvant therapy, surgical details and postoperative events.

ELIGIBILITY:
Inclusion Criteria:

* patients who received nipple sparing mastectomy and breast reconstruction from November 2018 to July 2022 from a single breast reconstruction surgeon.

Exclusion Criteria:

* patients failed to be examined for outcome evaluation will be excluded from the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who received nipple sparing mastectomy and breast reconstruction from November 2018 to July 2022 from a single breast reconstruction surgeon
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Successful | post-operative 7 days
  If the free flap transferred is successfully survived

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGungMH, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Wong AW, Kuo WL, Cheong DC, Tsai HP, Kao SW, Chen CF, Huang JJ. Six steps for a successful aesthetic free flap reconstruction after minimally invasive mastectomy: a retrospective case-control study. Int J Surg. 2024 Feb 1;110(2):645-653. doi: 10.1097/JS9.0000000000000871. PMID 38000051